CLINICAL TRIAL: NCT01409213
Title: Standardized Non-interventional Register Investigating the Daily Clinical Practice for the Treatment of Patients With Diabetes Mellitus Type 2 (SIRTA)
Brief Title: A Study of the Current Medical Practice and Outcomes in the Treatment of Type 2 Diabetes Mellitus in an Office Setting (MK-0431-199)
Acronym: SIRTA
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0431-199
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Results first posted 2012-01-23 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Enrolled Participants

SUMMARY:
The purpose of this study is to collect information of the risk profile of patients with type 2 diabetes mellitus, their treatment concerning meeting the guidelines for treatment of diabetic patients type 2 published by the Deutsche Diabetes Gesellschaft (DDG) on October 13, 2008

ELIGIBILITY:
Inclusion Criteria:

- Newly diagnosed with Type 2 diabetes in whom treatment with metformin in

the individual maximal tolerated dose (at least four weeks on stable dose) resulted in

HbA1c >6.5%

- No contraindication or intolerability to metformin

Exclusion Criteria:

- Currently being administered a combination therapy for the treatment of their Type 2 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with type 2 diabetes mellitus being treated in an office setting with metformin at the individual maximal tolerated dose (at least four weeks on stable dose) and had a resultant HbA1c >6.5% were selected for this study. The first five eligible participants per site with type 2 diabetes mellitus and treatment with metformin were to be enrolled.
Sampling Method: Probability Sample
Enrollment: 1523 (Actual)
Dates: Start 2009-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Full analysis set (FAS) consisted of 1522 participants; one participant was excluded from the FAS due to missing data at baseline.
Period: Overall Study
Arm/Group | All Enrolled Participants
Started | 1523
Completed | 1523
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Enrolled Participants: Full analysis set (FAS) consisted of 1522 participants; one participant was excluded from the FAS due to missing data at baseline.
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 1522
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (10.8)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 841
  Male | 680
  Missing | 1
Region of Enrollment [Number; unit: participants]
  Germany | 1522
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percent of glycosylated hemoglobin] — Population for this baseline characteristic consists of participants with available data, n=1519
  Percent of glycosylated hemoglobin | 7.4 (1.1)
Fasting blood glucose (FBG) [Mean (Standard Deviation); unit: mg/dL] — Population for this baseline characteristic consists of participants with available data, n=1366
  mg/dL | 146.9 (42.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline for Mean Hemoglobin A1c (HbA1C)
Description: Change from baseline was defined as mean HbA1c baseline value minus the mean HbA1c end of observation value.
Time Frame: Baseline and end of Observation (up to Month 6)
Population: Participants from the full analysis set with available data.
Measure: Mean (Standard Deviation); unit: Percent of glycosylated hemoglobin
Groups:
- All Enrolled Participants: All enrolled participants with available data.
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 1522
Percent of glycosylated hemoglobin
  End of observation, n=1483 | 6.9 (0.9)
  Change from baseline, n=1480 | -0.5 (1.0)

2. Primary Outcome: Change From Baseline for Mean Fasting Blood Glucose (FBG)
Description: Change from baseline was defined as mean FBG baseline value minus mean FBG end of observation value.
Time Frame: Baseline and end of Observation (up to Month 6)
Population: Participants from the full analysis set with available data.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 1346
mg/dL
  End of observation; n=1346 | 127.8 (34.7)
  Change from baseline, n=1244 | -18.6 (41.2)

ADVERSE EVENTS:
Description: Adverse events were not collected as part of this register. All adverse events occurring during the conduct of the register were to be reported to the pharmaceutical company responsible for the drug under which the participant experienced the adverse event.
Arm/Group | All Enrolled Participants
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No